CLINICAL TRIAL: NCT01968733
Title: A Randomized, Double-Blind, Multi-Center Study to Evaluate the Efficacy and Safety of Intravenous to Oral Solithromycin (CEM-101) Compared to Intravenous to Oral Moxifloxacin in the Treatment of Adult Patients With Community-Acquired Bacterial Pneumonia
Brief Title: Efficacy and Safety Study of Intravenous to Oral Solithromycin (CEM-101) Compared to Intravenous to Oral Moxifloxacin in Treatment of Patients With Community-Acquired Bacterial Pneumonia
Acronym: SOLITAIRE-IV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE01-301
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Community-acquired Bacterial Pneumonia
Keywords: Pneumonia; CABP; CAP; Macrolide
MeSH Terms: conditions — Pneumonia | interventions — solithromycin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxifloxacin (Active Comparator): Intravenous with the potential step-down to oral moxifloxacin
  Interventions: Drug: Moxifloxacin
- Solithromycin (Experimental): Intravenous with potential step-down to oral solithromycin
  Interventions: Drug: Solithromycin

INTERVENTIONS:
Drug: Solithromycin
  Other Names: CEM-101
  Arms: Solithromycin
Drug: Moxifloxacin
  Other Names: Avelox
  Arms: Moxifloxacin

SUMMARY:
This study will evaluate the safety and efficacy of an experimental antibiotic, solithromycin, in the treatment of adult patients with community-acquired pneumonia.

DETAILED DESCRIPTION:
Community-acquired bacterial pneumonia (CABP) is an acute infection of the pulmonary parenchyma with symptoms such as fever or hypothermia, chills, rigors, chest pain, and/or dyspnea. The widespread emergence of antibiotic resistant pathogens, including the macrolide-resistant Streptococcus pneumoniae, has resulted in a need for new and effective antibiotics that have activity against CABP pathogens. Solithromycin is a fourth generation macrolide antibiotic with excellent activity against resistant S. pneumoniae and other key typical and atypical bacterial respiratory pathogens. A completed Phase 2 study showed comparable efficacy to levofloxacin in adults with CABP.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years of age
* An acute onset of at least 3 of the following signs and symptoms (new or worsening):

  1. Cough
  2. Production of purulent sputum
  3. Shortness of breath (dyspnea)
  4. Chest pain due to pneumonia
* At least 1 of the following:

  1. Fever
  2. Hypothermia
  3. Presence of pulmonary rales and/or evidence of pulmonary consolidation
* PORT Risk Class II, III, or IV
* Presence of lobar, multilobar, or patchy parenchymal infiltrate(s) consistent with acute bacterial pneumonia on a pulmonary imaging study
* Not received any systemic antibiotics during the prior 7 days

Exclusion Criteria:

* Ventilator-associated pneumonia
* Known anatomical or pathological bronchial obstruction or a history of bronchiectasis or documented severe chronic obstructive pulmonary disease
* Hospitalization within 90 days or residence in a long-term care facility within 30 days prior to the onset of symptoms
* Fungal pneumonia
* Pneumocystis jiroveci pneumonia
* Aspiration pneumonia
* Other non-infectious causes of pulmonary infiltrates
* Primary or metastatic lung cancer
* Cystic fibrosis
* Active or suspected tuberculosis
* HIV or myasthenia gravis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 863 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Early clinical response rate in the Intent to Treat (ITT) population. | 72 [±12] hours after the first dose of study drug
  To determine noninferiority (NI) in early clinical response rate, in at least 2 of the following 4 cardinal symptoms: cough, shortness of breath, chest pain, and sputum production

SECONDARY OUTCOMES:
Early clinical response rate in the microITT population | 72 [±12] hours after the first dose of study drug
  To determine NI in early clinical response rate of intravenous to oral solithromycin compared to intravenous to oral moxifloxacin in the mITT population
Clinical success rates in the ITT and Clinically Evaluable (CE) populations | 5 to 10 days after the last dose of study drug
  To determine the overall clinical success rates of intravenous to oral solithromycin compared to moxifloxacin

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Jamieson, MD, Study Director — Melinta Therapeutics, Inc.
Locations (223):
- United States (56):
  - Mobile, Alabama
  - Little Rock, Arkansas
  - Chino, California
  - Glendale, California
  - Laguna Hills, California
  - Los Angeles, California
  - Pasadena, California
  - Sacramento, California
  - Sylmar, California
  - Torrance, California
  - Newark, Delaware
  - Bay Pines, Florida
  - DeLand, Florida
  - Doral, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - West Palm Beach, Florida
  - Augusta, Georgia
  - Blue Ridge, Georgia
  - Decatur, Georgia
  - Chicago, Illinois
  - Springfield, Illinois
  - Council Bluffs, Iowa
  - Hazard, Kentucky
  - Louisville, Kentucky
  - Owensboro, Kentucky
  - Lafayette, Louisiana
  - Shreveport, Louisiana
  - Detroit, Michigan
  - Farmington Hills, Michigan
  - Royal Oak, Michigan
  - Duluth, Minnesota
  - St Louis, Missouri
  - Butte, Montana
  - Newark, New Jersey
  - Somers Point, New Jersey
  - Buffalo, New York
  - Jamaica, New York
  - Johnson City, New York
  - New York, New York
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Lima, Ohio
  - Bethleham, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wyomissing, Pennsylvania
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Houston, Texas
  - Splendora, Texas
  - Charlottesville, Virginia
  - Spokane, Washington
- Argentina (11):
  - Caba, Buenos Aires
  - Florencia Varela, Buenos Aires
  - La Plata, Buenos Aires
  - Loma Hermosa, Buenos Aires
  - Mar del Plata, Buenos Aires
  - San Juan Bautista, Buenos Aires
  - Vicente López, Buenos Aires
  - Córdoba, Córdoba Province
  - Salta, Salta Province
  - Rosario, Santa Fe Province
  - San Miguel de Tucumán, Tucumán Province
- Bulgaria (8):
  - Kozloduy
  - Montana
  - Pernik
  - Rousse
  - Samokov
  - Sofia
  - Vidin
  - Vratsa
- Canada (8):
  - Edmonton, Alberta
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Chicoutimi, Quebec
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Sherbrooke, Quebec
- Chile (4):
  - Talca, Maule Region
  - Viña del Mar, Región de Valparaíso
  - Providencia, RM
  - Temuco
- Colombia (2):
  - Medellín, Antioquia
  - Cali, Valle del Cauca Department
- Georgia (3):
  - Batumi
  - Rustavi
  - Tbilisi
- Germany (7):
  - Bochum
  - Bonn
  - Dresden
  - Greifswald
  - Hanover
  - Lübeck
  - Rostock
- Guatemala (2):
  - Guatemala City, Departamento de Guatemala
  - Guatemala City
- Hungary (9):
  - Budapest
  - Debrecen
  - Győr
  - Kaposvár
  - Nagykanizsa
  - Nyíregyháza
  - Pécs
  - Székesfehérvár
  - Törökbálint
- Latvia (4):
  - Balvi
  - Daugavpils
  - Liepāja
  - Valmiera
- Malaysia (10):
  - Alor Star, Kedah
  - Kota Bharu, Kelantan
  - Cheras, Kuala Lumpur
  - Jalan Pahang, Kuala Lumpur
  - Malacca, Melaka
  - George Town, Pulau Pinang
  - Miri, Sarawak
  - Ampang, Selangor
  - Batu Caves, Selangor
  - Sungai Buloh, Selangor
- Netherlands (3):
  - Maastricht, Limburg
  - Breda, North Brabant
  - Utrecht, Utrecht
- Peru (13):
  - Ica, Ica
  - Miraflores, Lima 18
  - Cercado, Lima 1
  - San Juán de Miraflores, Lima 29
  - San Martín de Porres, Lima 31
  - San Miguel, Lima 32
  - Santiago de Surco, Lima 33
  - San Borja, Lima 41
  - Jesus Maria, Lima11
  - Lima Cercado, Lima1
  - Cercado, Lima
  - Iquitos, Loreto
  - Bellavista, Provincia Constitucional del Callao
- Philippines (5):
  - Lipa City, Batangas
  - EDSA Caloocan City, National Capital Region
  - Cebu City
  - Iloilo City
  - Quezon City
- Poland (6):
  - Chrzanów
  - Krakow
  - Lodz
  - Poznan
  - Warsaw
  - Wroclaw
- Romania (14):
  - Marghita, Bihor County
  - Bucharest, București
  - Cluj-Napoca, Cluj
  - Constanța, Constanța County
  - Craiova, Dolj
  - Bragadiru, Judet Ilfov
  - Suceava, Judetual Suceava
  - Ploieşti, Prahova
  - Bucharest, Sector 1
  - Bucharest, Sector 2
  - Bucharest, Sector 3
  - Bucharest, Sector 5
  - Suceava, Suceava
  - Timișoara, Timiș County
- Russia (8):
  - Barnaul
  - Chelyabinsk
  - Moscow
  - Novosibirsk
  - Penza
  - Saint Petersburg
  - Smolensk
  - Tomsk
- Serbia (4):
  - Belgrade
  - Kamenitz
  - Kragujevac
  - Niš
- Slovakia (3):
  - Kosice-Saca, Slovakia
  - Lučenec, Slovakia
  - Trebišov
- Slovenia (3):
  - Golnik
  - Ljubljana
  - Topolšica
- South Africa (7):
  - Benoni, Gauteng
  - Johannesburg, Gauteng
  - Krugersdorp, Gauteng
  - Newcastle, KwaZulu-Natal
  - Thabazimbi, Limpopo
  - Middleburg, Mpumalanga
  - Observatory, Western Cape
- South Korea (6):
  - Anyang-si, Gyenggi-do
  - Seoul, Gyenggi
  - Ansan-si, Gyeonggi-do
  - Goyang-si, Gyeonggi-do
  - Seoul, Gyeonggi-do
  - Jeonju, Jeollabuk-do
- Spain (9):
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Mataró, Barcelona
  - Granada, Granada
  - Madrid, Madrid
  - Torrejón de Ardoz, Madrid
  - Alicante
  - Barcelona
  - Madrid
- Taiwan (9):
  - Taichung, R.o. C.
  - Taipei, R.o. C.
  - Changhua Country
  - Hualien City
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Tainan
  - Taipei
- Ukraine (9):
  - Chernivtsi
  - Ivano Frakivsk
  - Kharkiv
  - Kherson
  - Kiev
  - Kremenchuk
  - Sumy
  - Vinnytsia
  - Zaporizhzhia

REFERENCES:
- [Derived] File TM Jr, Rewerska B, Vucinic-Mihailovic V, Gonong JRV, Das AF, Keedy K, Taylor D, Sheets A, Fernandes P, Oldach D, Jamieson BD. SOLITAIRE-IV: A Randomized, Double-Blind, Multicenter Study Comparing the Efficacy and Safety of Intravenous-to-Oral Solithromycin to Intravenous-to-Oral Moxifloxacin for Treatment of Community-Acquired Bacterial Pneumonia. Clin Infect Dis. 2016 Oct 15;63(8):1007-1016. doi: 10.1093/cid/ciw490. Epub 2016 Jul 22. PMID 27448679